CLINICAL TRIAL: NCT03085667
Title: Impact of Implantation of an LAA Occluder on ANP and BNP Level and Quality of Life
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Sven Möbius-Winkler, PI, University of Leipzig
Other Study IDs: SMW 05
Record Dates: First submitted 2016-10-25; First posted 2017-03-21 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation
Keywords: Left atrial appendage occluder; Watchman device; Atrial fibrillation; atrial natriureitc peptide; brain natriuretic peptide
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Closure of the LAA by several devices is a alternative therapy to oral anticoagulation in patients with Atrail fibrillation. Nothing is known about the acute influence of a device closure of the LAA on the secretion of ANB nad BNP hormones. Therefore aim of our study is to measure ANB and BNP levvels before and after Implantation of an LAA closure device.

DETAILED DESCRIPTION:
ANB and BNP levels are measured before, directly after and late after 24 h in central or periphereal venous blood from patients undergoing interventional LAA closure.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing LAA closure

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing left atrial appendage closure
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline atrial natriuretic Peptide (ANP) | 24 h post intervention
  comparison of ANP level pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sven Möbius-Winkler, MD, PhD, Principal Investigator — University of Leipzig
Locations (1):
- Heart Center Leipzig- University Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No